CLINICAL TRIAL: NCT03114449
Title: Auricular Acupuncture (AA) vs. Sham AA Procedure for Pain Control After Elective Knee Arthroplasty - a Randomized Controlled Trial
Brief Title: Auricular Acupuncture vs. Sham Procedure for Pain Control After Knee Arthroplasty
Acronym: AA_K-TEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Naemi-Wilke-Stift Guben Hospital - Anesthesia Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BB 102/11
Record Dates: First submitted 2017-04-03; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular acupuncture (Experimental): Auricular acupuncture (AA) with indwelling fixed needles at specific AA points
  Interventions: Device: Auricular acupuncture
- Sham auricular acupuncture (Sham Comparator): Sham auricular acupuncture with indwelling fixed needles at non- AA points
  Interventions: Device: Sham auricular acupuncture

INTERVENTIONS:
Device: Auricular acupuncture — Auricular acupuncture with indwelling fixed needles at specific AA points
  Arms: Auricular acupuncture
Device: Sham auricular acupuncture — Sham auricular acupuncture (AA) with indwelling fixed needles applied at non-AA points
  Arms: Sham auricular acupuncture

SUMMARY:
Aim of the study To investigate whether auricular acupuncture (AA) will reduce postoperative pain and analgesic requirement in comparison with sham AA in patients after elective knee arthroplasty

Design Prospective randomized controlled blinded clinical trial

Participants:

* Patients < 80 und > 50 years old
* scheduled for knee arthroplasty under general anesthesia with < 120 minutes duration
* Without previous opioid medication
* Able to give informed consent

Outcome measures

* Postoperative analgesic requirement
* Incidence of side effects
* Physiological parameters

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an American Society of Anesthesiologists physical status of I to III scheduled for elective knee arthroplasty under general anesthesia
2. Surgery time does not exceed 120 minutes
3. Patients without previous opioid medication
4. Patients ranged 50-80 years old
5. Patients who have given written informed consent

Exclusion Criteria:

1. Recidivist alcoholics
2. Local auricular skin infection
3. Age < 50 and > 80 years
4. Surgery time more than 120 minutes
5. Intraoperative complications (bleeding, required blood transfusion more than 6 units of packed cells, cardiovascular instability, required catecholamines)
6. Patients who consumed opioid medication at least 6 months before surgery
7. Patients with prosthetic or damaged cardiac valves, intracardiac and intravascular shunts, hypertrophic cardiomyopathy and mitral valve prolaps (risk of bacterial endocarditis according to guidelines of AHA)
8. Patients who are unable to understand the consent form
9. History of psychiatric disease

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Postoperative requirement of analgesic tilidine (measured in mg) | Six days following surgery
  Requirement of opioid analgesic tilidin

SECONDARY OUTCOMES:
Side effects of analgesics | Six days following surgery
  Incidence of nausea and vomiting
heart rate | 12 hours after surgery
  heart rate
blood pressure | 12 hours following surgery
  blood pressure
Patients' satisfaction with the treatment of postoperative pain using NRS-5 (where 1=excellent; 5=very bad) | 12 hours following surgery

IPD SHARING:
Plan to Share IPD: Undecided